CLINICAL TRIAL: NCT03544268
Title: Academic-Industrial Partnership for Translation of Acoustic Angiography
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: LCCC1748; 1R01CA189479-01 (NIH)
Record Dates: First submitted 2018-05-18; First posted 2018-06-01 (Actual); Results first posted 2022-04-01 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Signs and Symptoms
Keywords: ultrasound; breast; angiography
MeSH Terms: conditions — Signs and Symptoms | interventions — perflutren

STUDY DESIGN:
Intervention Model Description: Experimental: Acoustic Angiography
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Acoustic Angiography (Experimental): All clinical patients will be included in the experimental group.
  Interventions: Device: Acoustic Angiography; Drug: Definity
- Image Optimization (Experimental): In addition to clinical patients, 30 participants will be recruited to aid in optimizing the imaging parameters.
  Interventions: Device: Acoustic Angiography; Drug: Definity

INTERVENTIONS:
Device: Acoustic Angiography — Acoustic angiography imaging involves a research high frequency ultrasound scanner and a prototype transducer as well as conventional b-mode ultrasound to guide the location of the imaging. The conventional ultrasound will be conducted just prior to the acoustic angiography for localization. The imaging also requires administration of Definity ultrasound contrast agent.
  Acoustic angiography imaging will be performed by trained medical personnel using mild compression to eliminate motion. Total imaging time is estimated to be less than 15 minutes.
Drug: Definity — Baseline B-mode US will be performed to confirm the lesions being imaged (unless it is a subject with no lesions, then a basic B-mode US will be performed). Perflutren is a diagnostic drug that is intended to be used for contrast enhancement. The vial contains a clear, colorless, sterile, non-pyrogenic, hypertonic solution which is activated by mechanical agitation with Vialmix®.It will be dispensed in inactivated form to a study team member. The contrast agent will be activated just prior to administration (ideally to be used within 5 minutes of activation). Contrast agent Definity will be activated according to package insert instructions, including use of VialMix®, the device used to activate Definity. Administration will occur IV in coordination with staff trained specifically in contrast ultrasound imaging.The total imaging time is anticipated to be less than 30 minutes.

SUMMARY:
Purpose: The primary objective of this single arm study is to compare the sensitivity and specificity of acoustic angiography with traditional b-mode ultrasound in the distinction of malignant versus benign breast lesions. Secondary objectives include a comparison of area under the curve (AUC) for acoustic angiography versus b-mode ultrasound, and comparison of radiologist preference for the two imaging techniques for each of 3 lesion characteristics.

Participants: Sixty patients who are to have a clinical surgical breast biopsy based on results from pre-study standard of care (SOC) imaging will be recruited from the UNC Breast Clinic for participation in the study.

Procedures (methods): This is a one arm single center study of patients with suspicious breast lesions (BIRADS 4 or 5) from the UNC Breast Clinic that consent to undergo an acoustic angiography in conjunction with b-mode ultrasound prior to their scheduled biopsy.

DETAILED DESCRIPTION:
Increasing the sensitivity and specificity of diagnostic imaging in patients at high risk for breast cancer could provide substantial clinical benefit by improving diagnosis, preventing over-treatment, and reducing healthcare costs. Acoustic angiography is a new type of contrast enhanced ultrasound imaging which is specifically sensitive to microvascular structure and density. It evaluates tumor micro-vasculature and may provide a powerful prognostic tool for the diagnosis of breast cancer, and eventually for treatment evaluation.

Sixty patients who are to have a clinical surgical breast biopsy based on results from pre-study standard of care (SOC) imaging will be recruited from the UNC Breast Clinic for participation in the study. The primary objective of this single arm study is to compare the sensitivity and specificity of acoustic angiography with traditional b-mode ultrasound in the distinction of malignant versus benign breast lesions. Secondary objectives include a comparison of area under the curve (AUC) for acoustic angiography versus b-mode ultrasound, and comparison of radiologist preference for the two imaging techniques for each of 3 lesion characteristics.

ELIGIBILITY:
Inclusion Criteria

Subject must meet all of the inclusion criteria to participate in this study:

1. Women ≥18 years old
2. Patient had a diagnostic breast ultrasound study performed at UNC
3. Scheduled for a core needle or surgical breast biopsy of at least one breast lesion that is 2 cm or less in size and 3 cm in depth from the skin surface
4. Lesion visualized on ultrasound
5. Able to provide informed consent
6. Negative urine pregnancy test in women of child-bearing potential

Exclusion Criteria All subjects meeting any of the exclusion criteria at baseline will be excluded from study participation

1. Male (it is uncommon for men to present for imaging and the overwhelming majority of findings are non-cancerous and do not lead to biopsy; male breast cancer represents <1% of newly diagnosed breast cancer)
2. Institutionalized subject (prisoner or nursing home patient)
3. Critically ill or medically unstable and whose critical course during the observation period would be unpredictable (e.g., chronic obstructive pulmonary disease (COPD)
4. Sonographically visible breast lesion larger than 2cm or greater than 3cm in depth from the skin surface
5. Known hypersensitivity to sulfur hexafluoride or to any component of perflutren lipid (Definity®)
6. Active cardiac disease including any of the following:

   * Severe congestive heart failure (class IV in accordance with the classification of the New York Heart Association)
   * Unstable angina.
   * Severe arrhythmia (i.e. ventricular tachycardia, flutter fibrillation; ventricular premature complexes occurring close to the preceding T-wave, multifocal complexes).
   * Myocardial infarction within 14 days prior to the date of proposed Definity® administration.
   * Uncontrolled systemic hypertension (systolic blood pressure (BP) >150 mm Hg and/or diastolic BP >90 mm Hg despite optimal medical management).
7. Any woman who is pregnant or has reason to believe she is pregnant or any woman who is lactating (the possibility of pregnancy has to be excluded by negative urine β-HCG results, obtained within 24 hours before the perflutren lipid administration, or on the basis of patient history as defined by the UNC IRB SOP 4801 for child bearing potential)

Healthy Volunteers for Image Optimization

In addition to these clinical patients, 15 participants will be recruited to aid in optimizing the imaging parameters. These subjects must be willing to participate and able to provide written informed consent. However, these participants do not need to present any of the clinical indications as given for patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2021-05-25 (Actual); Study Completion 2021-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yueh Lee, MD, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Hospitals, Chapel Hill, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Acoustic Angiography: All clinical patients will be included in the experimental group.
  Acoustic Angiography: Acoustic angiography imaging involves a research high frequency ultrasound scanner and a prototype transducer as well as conventional b-mode ultrasound to guide the location of the imaging. The conventional ultrasound will be conducted just prior to the acoustic angiography for localization. The imaging also requires administration of Definity ultrasound contrast agent.
- Image Optimization: In addition to clinical patients, 30 participants will be recruited to aid in optimizing the imaging parameters.
  Acoustic Angiography: Acoustic angiography imaging involves a research high frequency ultrasound scanner and a prototype transducer as well as conventional b-mode ultrasound to guide the location of the imaging. The conventional ultrasound will be conducted just prior to the acoustic angiography for localization. The imaging also requires administration of Definity ultrasound contrast agent.
Period: Overall Study
Arm/Group | Acoustic Angiography | Image Optimization
Started | 5 | 15
Completed | 3 | 15
Not Completed | 2 | 0
Not completed — Did not meet full criteria for inclusion after enrollment | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acoustic Angiography | Image Optimization | Total
Number analyzed (Participants) | 5 | 15 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 15 | 20
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (4) | 26 (11) | 31 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 0 | 8 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 14 | 18
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 4 | 8 | 12
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 3 | 3
Region of Enrollment [Number; unit: participants]
  United States | 5 | 15 | 20

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity and Specificity
Description: To compare (using a reader study) the sensitivity and specificity of acoustic angiography to the sensitivity and specificity of conventional b-mode ultrasound in evaluation of breast lesions
Time Frame: 2 years
Population: The data were unable to be analyzed because we could not visualize the vessels to calculate this value. The system was unable to achieve the imaging resolution to visualize the vasculature.
Arm/Group | Acoustic Angiography | Image Optimization
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Area Under the Curve (AUC) of Acoustic Angiography
Description: To compare the area under the curve (AUC) of acoustic angiography to the AUC of the b-mode ultrasound To compare radiologist preference of acoustic angiography to conventional b-mode ultrasound for each lesion characteristic (shape, margins, and vascularity) Primary Endpoint Sensitivity and specificity for our study is defined as the ability of readers (radiologists) to use the acoustic angiography or b-mode ultrasound to distinguish between malignant and non-malignant breast lesions known to exist based on pathological results (the gold standard).
  The AUC of acoustic angiography compared to the AUC of b-mode ultrasound
Time Frame: 2 years
Population: as for outcome 1
Arm/Group | Acoustic Angiography | Image Optimization
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Radiologist Preference
Description: To compare radiologist preference of acoustic angiography to conventional b-mode ultrasound for each lesion characteristic (shape, margins and vascularity)
Time Frame: 2 years
Population: as for outcome 1
Arm/Group | Acoustic Angiography | Image Optimization
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Vessel Tortuosity (No Units)
Description: To quantify vessel tortuosity metrics for the acoustic angiograph images, and to use these metrics to develop a model for predicting malignancy (a model-based malignancy score)
Time Frame: 2 years
Population: as for outcome 1
Arm/Group | Acoustic Angiography | Image Optimization
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Model-based Malignancy Score (Arbitrary Units)
Description: To compare the model-based malignancy score to the acoustic angiography reader study
Time Frame: 2 years
Population: as for outcome 1
Arm/Group | Acoustic Angiography | Image Optimization
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 30 minutes post imaging
Arm/Group | Acoustic Angiography | Image Optimization
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/15
Other Adverse Events (participants affected / at risk) | 0/3 | 3/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Acoustic Angiography (N=3) | Image Optimization (N=15)
Flushing (Blood and lymphatic system disorders) | 0 | 3 — Flushing

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-08): https://cdn.clinicaltrials.gov/large-docs/68/NCT03544268/Prot_SAP_000.pdf